CLINICAL TRIAL: NCT03100370
Title: Effects of Combined Spinal Direct Current Stimulation on Upper Limb Recovery in Acquired Brain Injury (ABI)
Brief Title: Effects of Combined Spinal Direct Current Stimulation on Upper Limb Recovery in Acquired Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely due to COVID-19 pandemic.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Gerard Francisco, Professor, Physical Medicine and Rehabilitation, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-16-0237
Record Dates: First submitted 2016-11-23; First posted 2017-04-04 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Each participant will receive active anodal spinal stimulation, active cathodal spinal stimulation, and sham spinal stimulation. The order that each participant receives anodal, cathodal, and sham stimulation will be randomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- tsDCS-Anodal & robotic arm training (RAT), then tsDCS-Cathodal & RAT, then tsDCS-Sham & RAT (Experimental): anodal tsDCS over cervical spine, 2.5mA for 20 minutes
  Interventions: Device: tsDCS-Anodal Stimulation; Device: tsDCS-Cathodal Stimulation; Device: tsDCS-Sham Stimulation; Device: Robotic-assisted training of arm and hand functions
- tsDCS-Anodal & robotic arm training (RAT), then tsDCS-Sham & RAT, then tsDCS-Cathodal & RAT (Experimental): cathodal tsDCS over cervical spine, 2.5mA for 20 minutes
  Interventions: Device: tsDCS-Anodal Stimulation; Device: tsDCS-Cathodal Stimulation; Device: tsDCS-Sham Stimulation; Device: Robotic-assisted training of arm and hand functions
- tsDCS-Cathodal & robotic arm training (RAT), then tsDCS-Anodal & RAT, then tsDCS-Sham & RAT (Experimental): sham tsDCS over cervical spine, 2.5mA for 20 minutes
  Interventions: Device: tsDCS-Anodal Stimulation; Device: tsDCS-Cathodal Stimulation; Device: tsDCS-Sham Stimulation; Device: Robotic-assisted training of arm and hand functions
- tsDCS-Cathodal & robotic arm training (RAT), then tsDCS-Sham & RAT, then tsDCS-Anodal & RAT (Experimental)
  Interventions: Device: tsDCS-Anodal Stimulation; Device: tsDCS-Cathodal Stimulation; Device: tsDCS-Sham Stimulation; Device: Robotic-assisted training of arm and hand functions
- tsDCS-Sham & robotic arm training (RAT), then tsDCS-Anodal & RAT, then tsDCS- Cathodal & RAT (Experimental)
  Interventions: Device: tsDCS-Anodal Stimulation; Device: tsDCS-Cathodal Stimulation; Device: tsDCS-Sham Stimulation; Device: Robotic-assisted training of arm and hand functions
- tsDCS-Sham & robotic arm training (RAT), then tsDCS-Cathodal & RAT, then tsDCS-Anodal & RAT (Experimental)
  Interventions: Device: tsDCS-Anodal Stimulation; Device: tsDCS-Cathodal Stimulation; Device: tsDCS-Sham Stimulation; Device: Robotic-assisted training of arm and hand functions

INTERVENTIONS:
Device: tsDCS-Anodal Stimulation — 2.5mA anodal tsDCS over cervical spine for 20 minutes, five days a week, for two weeks. tsDCS electrodes will be placed over cervical spine and shoulder.
  Other Names: Transcutaneous Spinal Direct Current Stimulation
Device: tsDCS-Cathodal Stimulation — 2.5mA cathodal tsDCS over cervical spine for 20 minutes, five days a week, for two weeks. tsDCS electrodes will be placed over cervical spine and shoulder.
  Other Names: Transcutaneous Spinal Direct Current Stimulation
Device: tsDCS-Sham Stimulation — 2.5mA sham tsDCS over cervical spine for 20 minutes, five days a week, for two weeks. tsDCS electrodes will be placed over cervical spine and shoulder.
  Other Names: Transcutaneous Spinal Direct Current Stimulation
Device: Robotic-assisted training of arm and hand functions — 70 minutes of robotic-assisted training (RAT) of arm and hand functions will follow each of the tsDCS sessions, five days a week, for two weeks. Robotic-assisted training will be provided by using the MAHI Exo-II device.

SUMMARY:
This study will compare different polarities of transcutaneous spinal direct current stimulation combined with robotic-assisted arm training (RAT) in adults with acquired brain injury (ABI). Participants will receive 20 minutes of 2.5 milliamps (mA) anodal, cathodal, and sham transpinal direct current stimulation (tsDCS) over cervical spine combined with high intensity robotic-assisted arm training, five days a week, for 2 consecutive weeks.

DETAILED DESCRIPTION:
Acquired brain injury (ABI) is the leading cause of neurological disability in the United States and accounts for the poor physical health and the social dysfunction evident in survivors. Hemiparesis due to acquired brain injury is the primary cause of disability and arm paresis is perceived as the primary cause of disability by individuals who have suffered ABI because of the limitations it creates in performing activities of daily living (ADL). Rehabilitation of the impaired limb is essential for improving motor function after ABI, yet only 31% of ABI survivors receive outpatient rehabilitation. Therefore, effective therapy for upper-limb paresis must be addressed. Approximately 80% of all ABI survivors suffer from upper limb paresis and only 18% of these individuals gain full motor recovery with conventional treatments in the year following ABI.

The study will use cross-over, randomized, sham controlled, double-blinded design. Participants with subacute or chronic ABI will each be assigned to receive active anodal spinal stimulation, active cathodal spinal stimulation, and sham spinal stimulation for the same duration, and the order that each participant will receive anodal, cathodal, and sham stimulation will be randomized. In all the experiments participants will receive robotic assisted training for duration of 1.5 hours. The first 20 minutes of training will be coupled with spinal stimulation. Treatment will be administered at an intensity of 5 sessions per week for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Providing written informed consent prior to any study related procedures;
2. Age above 18;
3. Diagnosis of acquired brain injury at least for 6 month
4. No neuropsychiatric comorbidities
5. Not being involved in any specific exercise program (e.g., neuromuscular electrical stimulation (NMES), functional electrical stimulation (FES)) within the previous 3 months;
6. No planned alteration in upper-extremity therapy or medication for muscle tone during the course of the study;
7. Eligibility for standard upper-extremity rehabilitation at the time of enrollment (i.e., absence medical comorbidities that would prevent standard rehabilitation);
8. No condition (e.g., severe arthritis, extreme shoulder pain) that would interfere with valid administration of the measures or with interpreting motor testing;
9. No contraindications to tsDCS:

   * metal in the head between stimulation area
   * metal in the spine between stimulation area
   * implanted brain medical devices
10. No pregnancy;
11. No contraindications for Transcranial Magnetic Stimulation (TMS) and magnetic resonance imaging (MRI) based on TMS and MRI screening forms

Exclusion Criteria:

1. Uncontrolled epilepsy;
2. Any joint contracture or severe spasticity in the affected upper extremity, as measured by a Modified Ashworth Score > than 3 out of 4;
3. History of substance abuse;
4. Subject who cannot provide self-transportation to the study location

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Francisco, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The Institute for Rehabilitation and Research (TIRR) at Memorial Hermann, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuromodulation and Neural Interfaces Research Lab at Neurorecovery Research Center at The Institute for Research and Rehabilitation (TIRR) Memorial Hermann — https://med.uth.edu/pmr/research/neuromodulation-and-neural-interfaces-research/

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (2 Weeks)
Arm/Group | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Cathodal & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Anodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS- Cathodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Anodal & RAT
Started | 2 | 1 | 1 | 2 | 2 | 1
Completed | 2 | 1 | 1 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Washout (30 Days)
Arm/Group | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Cathodal & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Anodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS- Cathodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Anodal & RAT
Started | 2 | 1 | 1 | 1 | 2 | 1
Completed | 2 | 1 | 1 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Cathodal & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Anodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS- Cathodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Anodal & RAT
Started | 2 | 1 | 0 | 1 | 2 | 1
Completed | 2 | 1 | 0 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (30 Days)
Arm/Group | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Cathodal & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Anodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS- Cathodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Anodal & RAT
Started | 2 | 1 | 0 | 1 | 2 | 1
Completed | 2 | 1 | 0 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (2 Weeks)
Arm/Group | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Cathodal & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Anodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS- Cathodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Anodal & RAT
Started | 2 | 0 | 0 | 1 | 2 | 1
Completed | 2 | 0 | 0 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (30 Days)
Arm/Group | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Anodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Cathodal & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS-Sham & RAT | tsDCS-Cathodal & Robotic Arm Training (RAT), Then tsDCS-Sham & RAT, Then tsDCS-Anodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Anodal & RAT, Then tsDCS- Cathodal & RAT | tsDCS-Sham & Robotic Arm Training (RAT), Then tsDCS-Cathodal & RAT, Then tsDCS-Anodal & RAT
Started | 2 | 0 | 0 | 1 | 2 | 1
Completed | 2 | 0 | 0 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data were collected for all 9 participants that were enrolled. 8 of the 9 participants were assigned to and received any intervention.
Groups:
- All Study Participants: tsDCS-Anodal Stimulation & robotic-assisted training (RAT) of arm and hand functions: 2.5mA anodal tsDCS over cervical spine for 20 minutes followed by robotic-assisted training of arm and hand functions for 70 minutes, five days a week, for two weeks. tsDCS electrodes will be placed over cervical spine and shoulder. Robotic-assisted training will be provided by using the MAHI Exo-II device.
  tsDCS-Cathodal Stimulation & robotic-assisted training (RAT) of arm and hand functions: 2.5mA cathodal tsDCS over cervical spine for 20 minutes followed by robotic-assisted training of arm and hand functions for 70 minutes, five days a week, for two weeks. tsDCS electrodes will be placed over cervical spine and shoulder. Robotic-assisted training will be provided by using the MAHI Exo-II device.
  tsDCS-Sham Stimulation & robotic-assisted training (RAT) of arm and hand functions: 2.5mA sham tsDCS over cervical spine for 20 minutes followed by robotic-assisted training of arm and hand functions for 70 minutes, five days a week, for two weeks. tsDCS electrodes will be placed over cervical spine and shoulder. Robotic-assisted training will be provided by using the MAHI Exo-II device.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than One Race | 0
  Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Arm (FMA) Motor Score
Description: FMA is a stroke-specific, performance based impairment index. It quantitatively measures impairment based on Twitchell and Brunnstrom's concept of sequential stages of motor return in hemiplegic stroke patients. It uses an ordinal scale for scoring of 33 items for the upper limb component of the F-M scale (0:can not perform; 1:can perform partially; 2:can perform fully). Total range is 0-66, 0 being poor and 66 normal.
Time Frame: baseline
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- tsDCS- Anodal Stimulation & Robotic Arm Training (RAT): anodal tsDCS over cervical spine, 2.5mA for 20 minutes
  tsDCS-Anodal Stimulation: 2.5mA anodal tsDCS over cervical spine for 20 minutes followed by robotic-assisted training of arm and hand functions for 70 minutes, five days a week, for two weeks. tsDCS electrodes will be placed over cervical spine and shoulder. Robotic-assisted training will be provided by using the MAHI Exo-II device.
- tsDCS- Cathodal Stimulation & RAT: cathodal tsDCS over cervical spine, 2.5mA for 20 minutes
  tsDCS-Cathodal Stimulation: 2.5mA cathodal tsDCS over cervical spine for 20 minutes followed by robotic-assisted training of arm and hand functions for 70 minutes, five days a week, for two weeks. tsDCS electrodes will be placed over cervical spine and shoulder. Robotic-assisted training will be provided by using the MAHI Exo-II device.
- tsDCS- Sham Stimulation & RAT: sham tsDCS over cervical spine, 2.5mA for 20 minutes
  tsDCS-Sham Stimulation: 2.5mA sham tsDCS over cervical spine for 20 minutes followed by robotic-assisted training of arm and hand functions for 70 minutes, five days a week, for two weeks. tsDCS electrodes will be placed over cervical spine and shoulder. Robotic-assisted training will be provided by using the MAHI Exo-II device.
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 42 (13.8) | 40 (12.8) | 42.8 (12.7)

2. Primary Outcome: Fugl-Meyer Arm (FMA) Motor Score
Description: as for outcome 1
Time Frame: 2 weeks
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 43.1 (13.4) | 40.6 (13.4) | 44.2 (14.1)

3. Primary Outcome: Fugl-Meyer Arm (FMA) Motor Score
Description: as for outcome 1
Time Frame: 1 month
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 42.4 (14.7) | 42 (12.3) | 44.4 (13.5)

4. Secondary Outcome: Jebsen Taylor Hand Function Test (JTHFT)
Description: The JTHFT is a motor performance test and assesses the time needed to perform 7 everyday activities (for example, flipping cards and feeding). Score is reported as items completed per second.
Time Frame: Baseline
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: activities completed per second
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
activities completed per second | .22 (.2) | .17 (.2) | .23 (.2)

5. Secondary Outcome: Action Research Arm Test (ARAT)
Description: The ARAT is used to assess subject's ability to manipulate-lift-release objects horizontally and vertically, which differs in size, weight and shape. The test consists of 19 items divided into 4 sub-tests (grasp, grip, pinch, gross arm movement) and each item is rated on a 4-point scale. The possible total score ranges between 0-57. Higher scores indicate better performance.
Time Frame: Baseline
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 35.2 (22.8) | 34 (21.5) | 37.2 (23.1)

6. Secondary Outcome: Motor Activity Log (MAL)
Description: The MAL ranges from 0 to 5, with a higher score indicating greater ability to use the affected arm.
Time Frame: Baseline
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 1.99 (1.3) | 2.07 (1.4) | 2.15 (1.2)

7. Secondary Outcome: Pinch Strength
Description: A pinch gauge will be used to measure maximum pinch force.
Time Frame: Baseline
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: kg of force
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
kg of force | 11.2 (6.5) | 10.92 (11.8) | 9.4 (4.9)

8. Secondary Outcome: Quantitative Movement Measurement
Description: Robotic movement data will be used to quantitatively measure changes in movement smoothness
Time Frame: Change from baseline at 2 weeks and at 1 month
Population: Data were not collected for this outcome measure
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Adverse Effects Related to tsDCS
Description: Safety will be measured by questioning and observing participants at each treatment session. Adverse effects, such as skin redness etc. will be recorded.
Time Frame: Baseline
Population: Data were collected for 7 participants in each arm
Measure: Count of Participants; unit: Participants
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
Participants | 0 | 0 | 0

10. Secondary Outcome: Jebsen Taylor Hand Function Test (JTHFT)
Description: as for outcome 4
Time Frame: 2 weeks
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: activities completed per second
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
activities completed per second | .25 (.2) | .18 (.2) | .26 (.2)

11. Secondary Outcome: Jebsen Taylor Hand Function Test (JTHFT)
Description: as for outcome 4
Time Frame: 1 month
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: activities completed per second
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
activities completed per second | .25 (.2) | .2 (.2) | .22 (.2)

12. Secondary Outcome: Action Research Arm Test (ARAT)
Description: as for outcome 5
Time Frame: 2 weeks
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 36.7 (23.6) | 34.4 (21.6) | 40.1 (22.8)

13. Secondary Outcome: Action Research Arm Test (ARAT)
Description: as for outcome 5
Time Frame: 1 month
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 39.5 (22.7) | 35.1 (22.5) | 39 (23.6)

14. Secondary Outcome: Motor Activity Log (MAL)
Description: The MAL ranges from 0 to 5, with a higher score indicating greater ability to use the affected arm.
Time Frame: 2 weeks
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 2.17 (1.4) | 2.14 (1.4) | 2.07 (1.1)

15. Secondary Outcome: Motor Activity Log (MAL)
Description: The MAL ranges from 0 to 5, with a higher score indicating greater ability to use the affected arm.
Time Frame: 1 month
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | 2.34 (1.4) | 1.86 (1.6) | 2.2 (1.4)

16. Secondary Outcome: Number of Participants With Adverse Effects Related to tsDCS
Description: as for outcome 9
Time Frame: 2 weeks
Population: Data were collected for 7 participants in each arm
Measure: Count of Participants; unit: Participants
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
Participants | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Adverse Effects Related to tsDCS
Description: as for outcome 9
Time Frame: 1 month
Population: Data were collected for 7 participants in each arm
Measure: Count of Participants; unit: Participants
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
Participants | 0 | 0 | 0

18. Secondary Outcome: Pinch Strength
Description: A pinch gauge will be used to measure maximum pinch force.
Time Frame: 2 weeks
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: kg of force
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
kg of force | 12.1 (5.9) | 11.8 (3.9) | 10.9 (4.2)

19. Secondary Outcome: Pinch Strength
Description: A pinch gauge will be used to measure maximum pinch force.
Time Frame: 1 month
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: kg of force
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
kg of force | 10.4 (4.8) | 11.6 (3.6) | 9.5 (3.8)

20. Secondary Outcome: Grip Strength
Description: A grip dynamometer will be used to measure maximum gross grasp force.
Time Frame: baseline
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: kg of force
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
kg of force | 27.3 (17) | 22.1 (12.5) | 30.1 (18.3)

21. Secondary Outcome: Grip Strength
Description: A grip dynamometer will be used to measure maximum gross grasp force.
Time Frame: 2 weeks
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: kg of force
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
kg of force | 30.1 (19.1) | 21.8 (8.6) | 31.8 (15.8)

22. Secondary Outcome: Grip Strength
Description: A grip dynamometer will be used to measure maximum gross grasp force.
Time Frame: 1 month
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: kg of force
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
kg of force | 31.4 (18.7) | 22.5 (8.7) | 29.2 (6.0)

23. Secondary Outcome: Spasticity as Assessed by the Modified Ashworth Scale (MAS)
Description: This test measures spasticity in patients with lesions of the Central Nervous System by testing resistance to passive movement about a joint with varying degrees of velocity. Scores range from 0-4, with 0 indicating normal muscle tone and 4 indicating very high spasticity. The investigators will measure spasticity in the trained upper limb.
Time Frame: baseline
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | .2 (.2) | .4 (.4) | .3 (.3)

24. Secondary Outcome: Spasticity as Assessed by the Modified Ashworth Scale (MAS)
Description: as for outcome 23
Time Frame: 2 weeks
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | .2 (.3) | .3 (.2) | .3 (.2)

25. Secondary Outcome: Spasticity as Assessed by the Modified Ashworth Scale (MAS)
Description: as for outcome 23
Time Frame: 1 month
Population: Data were collected for 7 participants in each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 7 | 7 | 7
score on a scale | .05 (.09) | .2 (.2) | .3 (.3)

26. Secondary Outcome: Spinal Reflexes
Time Frame: Change from baseline at 2 weeks and at 1 month
Population: Data were not collected for this outcome measure
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Change in Strength of Selective Muscle Groups
Time Frame: Change from baseline at 2 weeks and at 1 month
Population: Data were not collected for this outcome measure
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Neurophysiologic Testing for Spinal Conductivity (SSEP)
Time Frame: Change from baseline at 2 weeks and at 1 month
Population: Data were not collected for this outcome measure
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | tsDCS- Anodal Stimulation & Robotic Arm Training (RAT) | tsDCS- Cathodal Stimulation & RAT | tsDCS- Sham Stimulation & RAT
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT03100370/Prot_SAP_000.pdf